CLINICAL TRIAL: NCT02615561
Title: Multicenter, Two-phase Exploratory Clinical Trial to Examine Efficacy and Safety After Open-label Topical Administration of a Medical Device (Bepanthen Itch Relief Cream) for Treatment of Acute Flare-ups Followed by Topical Administration of a New Cosmetic Bepanthen Product or a Cosmetic Comparator in a Parallel-group, Randomized, Investigator-blinded Care Phase for Skin Care in the Remission Phase in Infants With Mild Atopic Dermatitis
Brief Title: Curing Atopic Dermatits in Children With a Commerical Medical Device and Maintaining Healthy Skin by Using a New Cosmetic Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17534; 2015-003485-92 (EudraCT Number)
Record Dates: First submitted 2015-10-23; First posted 2015-11-26 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Dermatitis, Atopic
Keywords: Safety; Efficacy; Atopic dermatitis; Cosmetic products
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phase 1 (Cure phase) (Experimental): Efficacy and safety of the medical device Bepanthen Itch Relief Cream in children´s mild AD (responders will enter study phase 2)
  Interventions: Device: Bepanthen Itch Relief Cream: Phoenix 2 (Bepanthen Sensiderm, BAY207543)
- Phase 2 (Care phase) / Arm 1 (Experimental): Efficacy and safety of the new cosmetic Bepanthen test product in maintaining healthy skin in the remission phase after cure of children´s mild AD
  Interventions: Other: New cosmetic Bepanthen product: Pumpkin (BAY207543)
- Phase 2 (Care phase) / Arm 2 (Active Comparator): Efficacy and safety of Stelatopia (cosmetic comparator) in maintaining healthy skin in the remission phase after cure of children´s mild AD
  Interventions: Other: Stelatopia (cosmetic comparator)

INTERVENTIONS:
Device: Bepanthen Itch Relief Cream: Phoenix 2 (Bepanthen Sensiderm, BAY207543) — 2-3 times daily using multiples of Finger Tip Units (FTUs) depending on size of the area of the flares
  Arms: Phase 1 (Cure phase)
Other: New cosmetic Bepanthen product: Pumpkin (BAY207543) — Twice daily on the whole body; about 10 FTUs (i.e. 5g) per application depending on age of subject
  Arms: Phase 2 (Care phase) / Arm 1
Other: Stelatopia (cosmetic comparator) — Twice daily on the whole body; about 10 FTUs (i.e. 5g) per application depending on age of subject
  Arms: Phase 2 (Care phase) / Arm 2

SUMMARY:
1. Curing mild atopic dermatis in children with a commerical medical device (Bepanthen Itch Relief Cream).
2. Maintaining healthy skin by using a new cosmetic Bepanthen product or a commercially available cosmetic product

ELIGIBILITY:
Inclusion Criteria:

* Written parents' informed consent to have their child participate in the study and attend the study procedures and processes as outlined in the protocol
* Male or female babies/children aged between 1 month and 4 years
* Mild AD presenting a maximum SCORAD of 25 (at Screening and Baseline)
* Acute flare-up phase
* Local SCORAD ≥ 5 on the target area (at Screening and Baseline)
* Skin type I - IV according to Fitzpatrick

Exclusion Criteria:

* Any other skin disease at the target area that would interfere the clinical assessment in the opinion of the investigator
* Known allergies to any of the ingredients of the IMPs
* Any other adjuvant therapy for AD (UV therapy, probiotics, homeopathy etc.) within 30 days before Baseline as well as during the entire study
* Any use of another topical emollient or other established treatment for AD during Phase 1 (cure phase) and Phase 2 (care phase) at the site of flares (AD lesions). Exception are usual hygienic products in the nappy area

Ages: 1 Month to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 136 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-09-07 (Actual)

PRIMARY OUTCOMES:
Efficacy: SCORAD with included parameters "extent of disease/area affected" [%] as well as average intensity of pruritus and sleeplessness | up to 3 months
Efficacy: Local SCORAD including single symptoms erythema, edema/ papulation, excoriation, lichenification, oozing/crusts, dryness | up to 3 months
Efficacy: Quality of Life according to questionnaire | up to 3 months
Efficacy: Intensity of pruritus according to diary | up to 3 months
Efficacy: Intensity of sleeplessness according to diary | up to 3 months
Efficacy: Responder rate: No. of subjects with local SCORAD <5 (Phase 1, only) | up to 3 months
Efficacy: Time to flare-up (Phase 2, only) | up to 3 months
Efficacy: Percent of subjects with flare-up (Phase 2, only) | up to 3 months

SECONDARY OUTCOMES:
Safety: Number of adverse events (AE) | up to 3 months
Safety: physical examination | up to 3 months
  Weight and height
Safety: vital signs | up to 3 months
  Systolic and diastolic blood pressure, Heart rate
Safety: Local tolerability (by AE assessment) | up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Germany (14):
  - Karlsruhe, Baden-Wurttemberg
  - Kehl, Baden-Wurttemberg
  - Schwäbisch Hall, Baden-Wurttemberg
  - Welzheim, Baden-Wurttemberg
  - Altdorf B. Nürnberg, Bavaria
  - Neustadt / Aisch, Bavaria
  - Rosenheim, Bavaria
  - Bramsche, Lower Saxony
  - Bochum, North Rhine-Westphalia
  - Datteln, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Frankenthal, Rhineland-Palatinate
  - Neumünster, Schleswig-Holstein
  - Erfurt, Thuringia